CLINICAL TRIAL: NCT05924152
Title: A Phase 1, Open-label, One-sequence Crossover Study to Investigate the Effect of a Breast Cancer Resistance Protein Inhibitor on the Single-dose Pharmacokinetics of Adagrasib in Healthy Adult Subjects
Brief Title: A PK Study to Assess the Drug-drug Interaction of a BCRP Inhibitor on Adagrasib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 849-025
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy Adults
MeSH Terms: interventions — adagrasib; eltrombopag

STUDY DESIGN:
Intervention Model Description: One-sequence Crossover Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Active Comparator): Treatment A: A single oral dose of adagrasib 400 mg (2 × 200-mg tablets) on Day 1;
  Interventions: Drug: Adagrasib
- Treatment B (Active Comparator): Treatment B: A single oral dose of eltrombopag 75 mg
  (1 × 75-mg tablet) plus adagrasib 400 mg (2 × 200-mg tablets) on Day 8.
  Interventions: Drug: Eltrombopag + adagrasib

INTERVENTIONS:
Drug: Adagrasib — Adagrasib
  Arms: Treatment A
Drug: Eltrombopag + adagrasib — Eltrombopag + adagrasib
  Arms: Treatment B

SUMMARY:
A Phase 1, Open-label, One-sequence Crossover Study to Investigate the Effect of a Breast Cancer Resistance Protein Inhibitor on the Single-dose Pharmacokinetics of Adagrasib in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 60 years of age, inclusive, at Screening.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, or clinical laboratory evaluations at Screening and Check-in as assessed by the Investigator.
4. Females of childbearing potential will not be pregnant or lactating and must have a negative result on an approved pregnancy test at Screening and Check-in. Females of childbearing potential must agree to use contraception.
5. Male subjects must agree to use contraception.
6. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, thrombotic, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, any components of the investigational product (IP), or other substance (not including seasonal allergies).
3. History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (eg, uncontrolled nausea, vomiting, malabsorption syndrome).
4. Significant history or clinical manifestation of any hepatic disease, as determined by laboratory abnormalities.
5. History or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study.
6. Ventricular dysfunction or history of risk factors for Torsades de Pointes.
7. History of drug abuse within 2 years prior to Screening.
8. History of alcohol abuse within 12 months prior to Screening.
9. Positive serology test results for hepatitis B surface antigen, hepatitis C antibody, and/or human immunodeficiency virus (HIV) 1/2.
10. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in.
11. Use of any drugs or substances known or suspected to alter drug absorption, distribution, metabolism, or elimination.
12. Use or intend to use any prescription medications/products within 14 days prior to Check-in.
13. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations.
14. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days.
15. Subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUC (adagrasib) | Days 1 and 8
  Area under the plasma concentration-time curve (AUC) from time zero to infinity (AUC∞)
Pharmacokinetics - AUC (adagrasib) | Days 1 and 8
  AUC from time zero to the last quantifiable concentration (AUClast)
Pharmacokinetics - Cmax (adagrasib) | Days 1 and 8
  Maximum observed plasma concentration (Cmax)
Pharmacokinetics - Tmax (adagrasib) | Days 1 and 8
  Time to reach Cmax (tmax)
Pharmacokinetics - t1/2 (adagrasib) | Days 1 and 8
  Elimination half-life (t1/2)
Pharmacokinetics - CL/F (adagrasib) | Days 1 and 8
  Apparent total plasma clearance (CL/F)
Pharmacokinetics - Vz/F (adagrasib) | Days 1 and 8
  Apparent volume of distribution (Vz/F)

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 8 weeks from screening
  Incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea Clinical Research Unit Daytona Beach (Labcorp Clinical Research Unit Daytona Beach), Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No